CLINICAL TRIAL: NCT07299201
Title: Evaluation of the Efficiency of Proactive Telemedicine vs Face-to-Face Visits for Universal Access and Health Prevention in a Rural Primary Care Team: Randomized Non-Inferiority Clinical Trial
Brief Title: Proactive Telemedicine to Improve Healthcare Access and Prevention in Rural Primary Care (PTM)
Acronym: PTM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Catala de Salut (Other Government)
Responsible Party: Principal Investigator, Robert Panades Zafra, MD, Primary Care Physician, EAP Anoia Rural, Catalonia, Spain, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23/282-P
Record Dates: First submitted 2025-11-26; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Primary Health Care; Telemedicine; Face to Face Consultation; Health Care Access; Prevention; Quality of Life; Adverse Effects; Cardiovascular (CV) Risk; Behavior Change Interventions; Brief Intervention
Keywords: telemedicine; primary care access; non-inferiority trial; health behavior change; rural healthcare; preventive medicine; quality of life; proactive intervention

STUDY DESIGN:
Intervention Model Description: The study uses a two-arm parallel assignment model in which participants are randomly allocated to either the proactive telemedicine intervention or standard face-to-face care. Each participant remains in their assigned arm for the duration of the study, with no crossover.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Proactive Telemedicine (PTM) (Active Comparator): Participants receive proactive remote contact by telephone or secure electronic messaging. A standardized brief behavioral intervention is delivered at baseline, four months, and eight months, focusing on smoking status, alcohol consumption, Mediterranean diet adherence, and physical activity. The stage of behavioral change is assessed to tailor motivational strategies. Participants then enter an observational phase to monitor natural healthcare utilization.
  Interventions: Behavioral: Telemedicine Brief Behavioural Lifestyle Intervention
- Arm 2: Face-to-Face Consultation (Active Comparator): Participants attend in-person appointments at the health center at baseline, four months, and eight months. Each visit includes the same standardized behavioral intervention used in the PTM arm. Participants then enter an observational phase.
  Intervention: Face-to-Face Brief Behavioral Lifestyle Intervention
  Interventions: Behavioral: Face to face Brief Behavioural Lifestyle Intervention

INTERVENTIONS:
Behavioral: Telemedicine Brief Behavioural Lifestyle Intervention — Participants received proactive digital contact via phone or e-consultation. They underwent a brief behavioural intervention addressing modifiable lifestyle factors such as smoking, alcohol consumption, physical activity, and diet. Additionally, access to the rural primary healthcare system will also be measured.
  Arms: Arm 1: Proactive Telemedicine (PTM)
Behavioral: Face to face Brief Behavioural Lifestyle Intervention — Participants attend in-person visits where they undergo a brief behavioural intervention addressing modifiable lifestyle factors (smoking, alcohol, physical activity, diet). Additionally, access to the rural primary healthcare system is also measured.
  Arms: Arm 2: Face-to-Face Consultation

SUMMARY:
The study evaluates whether Proactive Telemedicine (PTM) can improve healthcare access for individuals who have not contacted their primary care team for at least one year, compared with face-to-face visits. PTM consists of brief, remote behavioral interventions addressing modifiable risk factors such as tobacco use, alcohol consumption (AUDIT-C: Alcohol Use Disorders Identification Test - Consumption), physical activity (IPAQ: International Physical Activity Questionnaire), and Mediterranean diet adherence (PREDIMED: Prevención con Dieta Mediterránea). PTM follows national preventive protocols including PAPPS (Programa de Actividades Preventivas y de Promoción de la Salud) and uses validated tools such as EuroQol-5D-5L (EQ-5D-5L) to measure healthcare accessibility and quality-of-life outcomes. This randomized non-inferiority trial aims to determine whether PTM is as effective and safe as traditional in-person consultations.

DETAILED DESCRIPTION:
Healthcare systems, particularly in rural and aging populations, face persistent challenges in ensuring equitable and universal access. Many individuals do not regularly engage with primary care services due to geographical, socioeconomic, organizational, or personal barriers. Digital health initiatives, including the World Health Organization's Global Strategy on Digital Health 2020-2025, highlight telemedicine as a key tool to improve accessibility and support preventive care.

Proactive Telemedicine (PTM) is a model in which primary care professionals initiate remote contact with individuals who have not interacted with their healthcare team for at least one year. The intervention uses synchronous (telephone) and asynchronous (secure messaging) communication to deliver brief behavioral counseling based on cognitive-behavioral and motivational interviewing principles. These interventions target modifiable lifestyle factors such as smoking, alcohol consumption, physical inactivity, and dietary patterns, and are aligned with national preventive care recommendations.

This randomized non-inferiority trial evaluates whether PTM provides accessibility, preventive impact, and user experience comparable to face-to-face consultations. The study examines whether proactively delivered telemedicine can serve as a scalable and acceptable strategy to increase engagement with primary care services in underserved rural areas. The information obtained will help determine the feasibility, effectiveness, and future implementation potential of PTM within broader healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Registered patients of EAP Anoia Rural
* Age ≥18 years
* No contact with the primary care team within the previous 12 months
* Able to provide informed consent (electronic or paper)

Exclusion Criteria:

* Proxy care (consulted by caregivers without patient present).
* Inability to communicate.
* Severe cognitive or psychiatric impairment.
* Advanced or palliative chronic conditions (MACA: Modelo de Atención Crónica Avanzada - Advanced Chronic Care Model).
* Outdated contact information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2026-03-16 (Estimated)

PRIMARY OUTCOMES:
Access to Primary Healthcare | 12-month post-intervention
  Proportion of participants who initiate any contact with primary care during the 12-month post-intervention observation period.
  Unit of Measure: Proportion (%)
Health-Related Quality of Life, EuroQol-5D-5L (EQ-5D-5L) | Baseline, 4 months, 8 months
  Change in quality-of-life score measured using the EuroQol-5D-5L instrument. Unit of Measure: Index score (0-1)

SECONDARY OUTCOMES:
Smoking Status | Baseline, 4 months, 8 months
  Change in categorical smoking status (smoker/non-smoker). Unit of Measure: Categorical.
Alcohol Consumption (AUDIT-C) | Baseline, 4 months, 8 months
  Change in score on the AUDIT-C questionnaire. Unit of Measure: Score (0-12).
Mediterranean Diet Adherence (PREDIMED) | Baseline, 4 months, 8 months
  Change in PREDIMED score. Unit of Measure: Score (0-14).
Physical Activity (IPAQ) | Baseline, 4 months, 8 months
  Change in physical activity level. Unit of Measure: MET-minutes/week (Low: <600, Moderate: 600-2999, High: ≥3000)
Stage of Behavioral Change | Baseline, 4 months, 8 months
  Change in stage of change using transtheoretical model. Unit of Measure: Categorical (precontemplation, contemplation, preparation, action, maintenance, relapse)
Coronary Risk (REGICOR Score) | Baseline and 8 months
  Change in 10-year coronary risk percentage calculated using REGICOR function. Unit of Measure: Percentage (%),
Morbidity Assessment | Baseline to 8 months
  Change in number and type of chronic conditions documented in electronic health records (ECAP).
  Unit of Measure: Count of conditions.
Patient Satisfaction | At 8 months
  Satisfaction score using validated telemedicine satisfaction survey (adapted from Tovar-Martínez et al.).
  Unit of Measure: Score (Likert scale).
Adverse Effects | Baseline to 8 months
  Number of intervention-related adverse events. Unit of Measure: Count

CONTACTS AND LOCATIONS:
Overall Officials: Josep Vidal Alaball, PhD, Study Director — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina; Robert Panadés Zafra, MD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- EAP Anoia rural. Gerència d'Atenció Primària i a la comunitària Penedès. Institut Català de la Salut. Departament de Salut. Generalitat de Catalunya, Igualada, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osman S, Churruca K, Ellis LA, Luo D, Braithwaite J. The Unintended Consequences of Telehealth in Australia: Critical Interpretive Synthesis. J Med Internet Res. 2024 Aug 27;26:e57848. doi: 10.2196/57848. PMID 39190446
- [Background] Goncalves-Bradley DC, J Maria AR, Ricci-Cabello I, Villanueva G, Fonhus MS, Glenton C, Lewin S, Henschke N, Buckley BS, Mehl GL, Tamrat T, Shepperd S. Mobile technologies to support healthcare provider to healthcare provider communication and management of care. Cochrane Database Syst Rev. 2020 Aug 18;8(8):CD012927. doi: 10.1002/14651858.CD012927.pub2. PMID 32813281
- [Background] Direcció General de Planificació en Salut. Document tècnic de l'Enquesta de salut de Catalunya 2021. Barcelona; 2022 Jun.
- [Background] Flodgren G, Rachas A, Farmer AJ, Inzitari M, Shepperd S. Interactive telemedicine: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2015 Sep 7;2015(9):CD002098. doi: 10.1002/14651858.CD002098.pub2. PMID 26343551
- [Background] MSSSI, 2015. Consejo integral en estilo de vida en atención primaria, vinculado con recursos comunitarios en población adulta. Estrategia de Promoción de la Salud y Prevención en el SNS. Ministerio de Sanidad, Servicios Sociales e Igualdad. Madrid; 2015.
- [Background] Cordoba Garcia R, Camarelles Guillem F. [Screening and brief intervention on alcohol consumption]. Aten Primaria. 2022 Jul;54(7):102349. doi: 10.1016/j.aprim.2022.102349. Epub 2022 May 9. Spanish. PMID 35550977
- [Background] Rosembaun A, Rojas P, Rodriguez MV, Barticevic N, Rivera Mercado S. Brief interventions to promote behavioral change in primary care settings, a review of their effectiveness for smoking, alcohol and physical inactivity. Medwave. 2018 Jan 29;18(1):e7148. doi: 10.5867/medwave.2018.01.7148. English, Spanish. PMID 29385118
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] McGovern L, Miller G, Hughes-Cromwick P. The Relative Contribution of Multiple Determinants to Health Outcomes. Researchers continue to study the many interconnected factors that affect people's health. Heal Policy Br. 2014 Aug 21;1-9.
- [Background] Stringhini S, Sabia S, Shipley M, Brunner E, Nabi H, Kivimaki M, Singh-Manoux A. Association of socioeconomic position with health behaviors and mortality. JAMA. 2010 Mar 24;303(12):1159-66. doi: 10.1001/jama.2010.297. PMID 20332401
- [Background] Littenberg B, Strauss K, MacLean CD, Troy AR. The use of insulin declines as patients live farther from their source of care: results of a survey of adults with type 2 diabetes. BMC Public Health. 2006 Jul 27;6:198. doi: 10.1186/1471-2458-6-198. PMID 16872541
- [Background] Kruzich JM, Jivanjee P, Robinson A, Friesen BJ. Family caregivers' perceptions of barriers to and supports of participation in their children's out-of-home treatment. Psychiatr Serv. 2003 Nov;54(11):1513-8. doi: 10.1176/appi.ps.54.11.1513. PMID 14600311
- [Background] Equip ESCA del Departament de Salut. Document tècnic de l ' Enquesta de salut de Catalunya (ESCA). Barcelona; 2016.
- [Background] Sandoval B, Martínez C, Llobet V, Belmonte T, Vilarasau R, Sandoval NB, et al. Validación de la versión en español del cuestionario PCAS para evaluar la atención primaria de salud. Rev Panam Salud Publica;31(1),ene 2012. 2012;31(1):2012.
- [Background] Ramsay J, Campbell JL, Schroter S, Green J, Roland M. The General Practice Assessment Survey (GPAS): tests of data quality and measurement properties. Fam Pract. 2000 Oct;17(5):372-9. doi: 10.1093/fampra/17.5.372. PMID 11021894
- [Background] Bower P, Roland M, Campbell J, Mead N. Setting standards based on patients' views on access and continuity: secondary analysis of data from the general practice assessment survey. BMJ. 2003 Feb 1;326(7383):258. doi: 10.1136/bmj.326.7383.258. PMID 12560279
- [Background] Sans-Corrales M, Pujol-Ribera E, Gene-Badia J, Pasarin-Rua MI, Iglesias-Perez B, Casajuana-Brunet J. Family medicine attributes related to satisfaction, health and costs. Fam Pract. 2006 Jun;23(3):308-16. doi: 10.1093/fampra/cmi112. Epub 2006 Feb 3. PMID 16461452
- [Background] Bashshur RL, Reardon TG, Shannon GW. Telemedicine: a new health care delivery system. Annu Rev Public Health. 2000;21:613-37. doi: 10.1146/annurev.publhealth.21.1.613. PMID 10884967
- [Background] Rabanales Sotos J, Párraga Martínez I, López-Torres Hidalgo J, Andrés Pretel F, Navarro Bravo B. Tecnologías de la Información y las Comunicaciones: Telemedicina. Rev Clin Med Fam. 2011 Feb;4(1):42-8.
- [Background] PAHO. Framework for the Implementation of a Telemedicine Service. Pan American Organization, World Health Organization. 2016. p. 67
- [Background] Barbosa W, Zhou K, Waddell E, Myers T, Dorsey ER. Improving Access to Care: Telemedicine Across Medical Domains. Annu Rev Public Health. 2021 Apr 1;42:463-481. doi: 10.1146/annurev-publhealth-090519-093711. PMID 33798406
- [Background] Ekeland AG, Bowes A, Flottorp S. Effectiveness of telemedicine: a systematic review of reviews. Int J Med Inform. 2010 Nov;79(11):736-71. doi: 10.1016/j.ijmedinf.2010.08.006. PMID 20884286
- [Background] Dorsey ER, Topol EJ. State of Telehealth. N Engl J Med. 2016 Jul 14;375(2):154-61. doi: 10.1056/NEJMra1601705. No abstract available. PMID 27410924
- [Background] Organización Mundial de la Salud. La OMS publica las primeras directrices sobre intervenciones de salud digital. Ginebra; 2019.
- [Background] World Health Organization. Proyecto de estrategia mundial sobre salud digital 2020-2025. 2020;42.
- [Background] Tovar-Martinez JI, Romero-Ibarguengoitia ME, Elvira Torres-Almaguer C. Development and Validation of an Instrument in Spanish to Evaluate Patient Satisfaction in Telemedicine Consultation During COVID-19 Pandemic. Telemed J E Health. 2022 May;28(5):736-742. doi: 10.1089/tmj.2021.0320. Epub 2021 Sep 9. PMID 34515522
- See also: Background resource on access to health services as a social determinant of health, from Healthy People 2030. — https://odphp.health.gov/healthypeople/priority-areas/social-determinants-health/literature-summaries/access-health-services